CLINICAL TRIAL: NCT01822002
Title: Randomized Controlled Trials for Treatment of Benign Paroxysmal Positional Vertigo
Brief Title: Treatment of Posterior Canal Type of Benign Paroxysmal Positional Vertigo
Acronym: PC-BPPV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chonbuk National University (Other)
Responsible Party: Principal Investigator, Sun-Young Oh, Professor, Chonbuk National University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Treatment of PC-BPPV
Record Dates: First submitted 2013-03-25; First posted 2013-04-01 (Estimated); Last update posted 2013-04-01 (Estimated); Status verified 2013-03

CONDITIONS: Benign Paroxysmal Positional Vertigo (BPPV)
Keywords: Vertigo; Nystagmus; BPPV = benign paroxysmal positional vertigo; Treatment outcome
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo; Vertigo; Nystagmus, Pathologic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Canalith repositionig maneuver; Epley maneuver group (Active Comparator): Patients with PC-BPPV will be randomly assigned to Epley maneuver or Semont maneuver.
  Interventions: Procedure: Canalith repositioning maneuver
- Canalith repositioning maneuver : Semont maneuver group (Active Comparator): Patients with PC-BPPV will be randomly assigned to Epley maneuver or Semont maneuver group.
  Interventions: Procedure: Canalith repositioning maneuver

INTERVENTIONS:
Procedure: Canalith repositioning maneuver
  Other Names: Epley maneuver; Semont maneuver

SUMMARY:
To determine the immediate therapeutic efficacies of canalith repositioning maneuvers in each type of BPPV (posterior canal type, apogeotropic horizontal canal type and geotropic horizontal canal type).

DETAILED DESCRIPTION:
In nationwide 10 Dizziness Clinics of Korea, consecutive patients with each type of BPPV are randomized to each repositioning maneuver.

For posterior canal type of BPPV (PC-BPPV), patinets are randomized into modified Epley maneuver and Semont maneuver.

Subjects Consecutive patients with a diagnosis of PC-BPPV are recruited from nationwide 10 Dizziness Clinics in Korea. The inclusion criteria for this study were (1) a history of positional vertigo, (2) direction-changing positional nystagmus appropriate for each type of BPPV, and (3) absence of identifiable central nervous system disorders that could explain the positional vertigo and nystagmus. To exclude the patients with nystagmus from central pathologies, all patients also will receive neurotological examinations including spontaneous and gaze-evoked (GEN) nystagmus, horizontal and vertical smooth pursuit and saccades, limb ataxia, and balance function in addition to routine neurological examinations. Even in patients with isolated vertigo, those with central ocular motor signs, limb ataxia, and severe imbalance will be arranged for MRIs.

Diagnostic procedure To induce positional nystagmus, the patients lied supine from sitting (lying-down nystagmus) and turned their heads to either side while in supine (head-turning nystagmus). Then the patients were moved from a supine to sitting position and the head was bent down (head-bending nystagmus). Patients were also subjected to right and left Hallpike maneuvers and straight head hanging test to exclude BPPV involving the posterior or anterior canal.

Study design and Randomization The investigators attempt to determine the immediate therapeutic efficacies of Epley maneuver and Semont maneuver for PC-BPPV, repeated barbecue rotation maneuver and Gufoni maneuver after barbecue rotatio maneuver for geotropic HC-BPPV, and repeated Gufoni maneuver and head-shaking maneuvers after Gufoni maneuver in apogeotropic HC-BPPV by adopting a prospective randomized controlled study design.

Based on the data from the pilot study, the investigators estimated the proportion of immediate resolution would be 60-70% in the repositioning groups. By adopting 0.9 power to detect a significant difference (p=0.05, two-sided) and a drop rate of 5%, 200 patients of each type of BPPV will be required for each treatment arm.

The immediate treatment response will be determined by participating neurologists in each clinic without knowing the maneuver applied to each patient from 30 minutes to one hour after initial maneuver. The absence of both vertigo and nystagmus will be required to determine a resolution. When the patient still show positioning nystagmus or vertigo, the patient will be received the another maneuver at each protocol arm.

ELIGIBILITY:
Inclusion Criteria:

1. a history of positional vertigo
2. upbeating-torsional nystagmus in Dix-Hallpike maneuver
3. absence of identifiable central nervous system disorders that could explain the positional vertigo and nystagmus.

Exclusion Criteria:

(1) Patients with positive neurotological examinations including spontaneous and gaze-evoked (GEN) nystagmus, horizontal and vertical smooth pursuit and saccades, limb ataxia, and balance function in addition to routine neurological examinations.

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
efficacy of repositioning maneuvers for treating PC-BPPV | 2hr
  The immediate treatment response will be determined by participating neurologists in each clinic without knowing the maneuver applied to each patient from 30 minutes to one hour after initial maneuver. The absence of both vertigo and nystagmus will be required to determine a resolution.

CONTACTS AND LOCATIONS:
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea

REFERENCES:
- [Derived] Oh SY, Kim JS, Choi KD, Park JY, Jeong SH, Lee SH, Lee HS, Yang TH, Kim HJ. Switch to Semont maneuver is no better than repetition of Epley maneuver in treating refractory BPPV. J Neurol. 2017 Sep;264(9):1892-1898. doi: 10.1007/s00415-017-8580-2. Epub 2017 Jul 28. PMID 28755307